CLINICAL TRIAL: NCT02076087
Title: Immune Characterization of Subcutaneous Adipose Tissue
Acronym: ATI
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-02113
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Determine Immune Cell Types in Subcutaneous Adipose Tissue
Keywords: Subcutaneous adipose tissue; Lipectomy
MeSH Terms: interventions — Lipectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum and plasma samples will be obtained Abdominal and thigh subcutaneous adipose tissue obtained during surgery
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Normal Weight (BMI: 18.5-24.9 kg/m²): Liposuction/lipectomy
  Interventions: Procedure: Liposuction/lipectomy
- Overweight (BMI: 25.0-29.9 kg/m²): Liposuction/lipectomy
  Interventions: Procedure: Liposuction/lipectomy
- Obese (BMI: >30.0kg/m²): Liposuction/lipectomy
  Interventions: Procedure: Liposuction/lipectomy

INTERVENTIONS:
Procedure: Liposuction/lipectomy — Subcutaneous adipose tissue will be obtained from liposuction/lipectomy to determine the types of immune cells

SUMMARY:
The overall goal of this proposal is to characterize the immune cell profile of subcutaneous abdominal adipose tissue in lean, overweight, obese and lipedema adults, and to evaluate potential associations between different adipose tissue immune cell types and metabolic profile.

ELIGIBILITY:
Inclusion Criteria:

* Women of all races and ethnicity
* Age between 18 and 65 years
* Body Mass Index (BMI) ≥ 18.5 kg/m²
* Weight stable (+/- 3% during the last 2 months before enrollment)
* Women already scheduled for above mentioned procedures

Exclusion Criteria:

* Diabetes Mellitus
* Recent (<5 years) history of cancer (except in situ ductal breast carcinoma)
* Chemotherapy and/or radiation therapy within 4 months before enrollment
* Immune system diseases (i.e., autoimmune disorders, acquired immunodeficiency syndrome)
* Pregnant or breastfeeding
* Take any medication that might affect immune function
* Severe organ dysfunction
* BMI <18.5 kg/m² or size of each breast is >600 grams, if scheduled for bilateral breast reconstruction

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 women already scheduled to undergo liposcution/lipectomy procedure for breast reconstruction associated with prophylactic mastectomy or mastectomy for in situ ductal breast corcinoma, cosmetic surgery, or abdominal lipectomy for severe obesity at either Barnes-Jewish Hospital or Barnes-Jewish West County Hospital. Subjects of all races and ethnicity, with a body mass index (BMI) greater than or equal to 18.5 kg/m² and between the ages of 18 and 65 years of age will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Determine the types of immune cells and the relative prevalence of each type and sub-type, in subcutaneous adipose tissue of normal weight, overweight, obese and lipedema adults. | intraoperative

SECONDARY OUTCOMES:
Determine the relationships among specific types and subtypes of immune cells, adiposity and cardiometabolic risk. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States